CLINICAL TRIAL: NCT01588665
Title: Relative Contributions of Red Cell Catabolism and Dietary Absorption to Fetal Iron Accretion During Pregnancy
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 1203002861
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Iron Deficiency
Keywords: pregnancy; stable isotopes; red blood cell catabolism
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A total of 45 mL maternal blood sample is collected at five study visits during pregnancy
  * At delivery, an additional 10 mL maternal blood sample, a 30 mL cord blood, and the placenta are collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women and pregnant adolescents

SUMMARY:
The two specific aims of this study are 1) to assess the relative contributions of two major maternal iron sources (i.e. dietary iron intake and red cell catabolism) at supplying iron to the fetus, and 2) to determine the impact of maternal and fetal iron status on placental transfer of these two iron sources in pregnant women and adolescents during the last trimester of pregnancy.

DETAILED DESCRIPTION:
Pregnant women and adolescents (n=24) will be recruited when entering prenatal care. They will be invited to participate in a longitudinal study comparing the relative contribution of the two major maternal iron sources, i.e. maternal dietary iron intake and maternal red blood cell iron recycling, to fetal iron accretion during pregnancy. At about 15 weeks of gestation, participants will consume an oral dose of a stable iron isotope (57Fe as ferrous sulfate) to enrich their red blood cells (RBCs) with 57Fe. Maternal blood samples will be collected at 4 times during pregnancy to monitor changes in blood 57Fe concentrations. In the third trimester of pregnancy, women will consume a dose of a different iron isotope (58Fe as ferrous sulfate) as dietary nonheme iron. Cord blood samples and placental tissue will be obtained at delivery to determine how much of the dietary iron (58Fe) and RBC iron (57Fe) was transferred to the fetus and how much of each isotope was retained in the placenta. Placenta tissue samples will also be used to assess placental expression of iron transporters in relation to the amount of each iron isotopes transferred to the fetus. Circulating iron status indicators and regulators will be measured in all maternal and cord blood samples to examine the effect of iron status on placental transfer of iron derived from the diet vs. RBC during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Non-smoker
* No pre-existing medical complications (such as HIV-infection, eating disorders, hemoglobinopathies, malabsorption diseases, steroid use, substance abuse history, or taking medications known to influence iron homeostasis)

Exclusion Criteria:

* Complicated pregnancy (including gestational diabetes, pregnancy-induced hypertension, or preeclampsia)
* Individuals been previously treated for lead exposure, or those that have been identified as having elevated blood lead concentrations during childhood, will be excluded from the study

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women and pregnant adolescents from Rochester, NY (n=24)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Transfer of iron to the fetus | The delivery study will be undertaken over a 24 h period

SECONDARY OUTCOMES:
Maternal and neonatal micronutrient status | Participants will be followed over the course of the pregnancy for an average of 28 weeks. The delivery study will be undertaken over a 24 h period.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O'Brien, PhD, Principal Investigator — Cornell University
Locations (1):
- Highland Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No